CLINICAL TRIAL: NCT02820909
Title: Interest of the Ultrasound Guidance for the Laying of Femoral Arterial and Venous Catheters in Intensive Care Unit: A Controlled, Randomized Trial: The ECHOGUIDE Study
Brief Title: Interest of the Ultrasound Guidance for the Laying of Femoral Arterial and Venous Catheters in Intensive Care Unit
Acronym: ECHOGUIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 69HCL16_0403
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Severely Traumatized Patients in Emergency Wards
Keywords: ultrasound guidance; emergency wards; arterial and venous catheters; femoral; complications
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound guidance (Experimental): 46 patients in the experimental ultrasound group
  Interventions: Procedure: venous and arterial catheter set-up using ultrasound guidance
- Anatomical guidance (Active Comparator): 46 patients in the anatomical group
  Interventions: Procedure: Anatomical guidance.

INTERVENTIONS:
Procedure: venous and arterial catheter set-up using ultrasound guidance — The insertion of the venous and arterial catheter will be done using ultrasound guidance. Vein and artery will be identified in cross section. In case of anatomical difficulties, complications of puncture with anatomical landmarks, or if installation time is greater than > 5 minutes, an intra-osseous catheter will be put in place to avoid delaying of treatment according to the current practice of the intensive care unit.
  Arms: Ultrasound guidance
Procedure: Anatomical guidance. — In the anatomical group, catheter will be inserted using, as it is currently done in intensive care unit, anatomic landmarks. If catheterization according to the anatomic method is considered too difficult (> 3 punctures), a conversion to ultrasound guidance will be done.
  In case of anatomical difficulties, complications of puncture with anatomical landmarks, or if installation time is greater than > 5 minutes, an intra-osseous catheter will be put in place to avoid delaying of treatment according to the current practice of the intensive care unit.
  Arms: Anatomical guidance

SUMMARY:
The femoral approach is the preferred vascular access for the set-up of emergency catheters in severely traumatized patient. This location combines simplicity and speed of installation, it allows the simultaneous set-up of arterial and venous catheters, and is a provider of few complications and failures.

The ultrasound guidance has greatly reduced installation times, failures and complications related to the set-up of central venous catheter. This was amply demonstrated in the internal jugular and subclavian site outside of extreme emergency situations (Fragou M et al 2011, Farrell J et al 1997, Karakistos et al 2006). The benefit of ultrasound guidance for the set-up of arterial and venous catheters in the femoral emergency has not been evaluated in terms of reduction in complications.

Then the main objective of this study is to demonstrate that the ultrasound guidance reduces early complications related to the set-up of arterial and venous catheters in the femoral emergency, among severely traumatized patient compared to the reference anatomical technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Included in intensive care unit for severe trauma
* Need for implementation of femoral arterial and venous catheters in accordance with the practices of the service.
* Agreed to participate
* Affiliation to national security

Exclusion Criteria:

* Contraindication to the set-up of vascular access in femoral position (femoral Scarpa wound, aortic dissection)
* Local infection
* Hypothermia <32°C
* Need for implementation of arterial catheter only
* Need for implementation of venous catheter only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Proportion of complications 1 week after catheter set-up. | 1 week.
  The primary end point is the proportion of patients with a complication one week after arterial and venous catheter set-up.
  Complications will be defined as follows:
  * mechanical immediate complications (hematoma, bleeding, dysfunction or non-function of the catheter, or aberrant course subcutaneous catheter)
  * Mechanical complications remote installation catheters (arteriovenous fistula, pseudoaneurysm), thrombotic complications.
  Vascular assessment will be conducted by an angiologist, using doppler ultrasound of the femoral vessels. Assessment will be made blind from the use of ultrasound guidance during installation.

SECONDARY OUTCOMES:
Cannulation time between the 2 groups | the day of surgery (Day 1)
  Comparison of cannulation mean time between the ultrasound guidance group and anatomical guidance group.
  Cannulation time is defined as the time in seconds, from the first contact between the needle and the skin, and when the two guide wires are inserted into the vessels (artery and vein).
total catheter set-up time between the 2 groups | the day of intervention (Day 1)
  Comparison of total catheter set-up mean time between the ultrasound guidance group and anatomical guidance group.
  Total exposure time of the catheter is defined as the time, in seconds, from the first contact between the needle and the skin, and when the dressing is applied to both catheters in place and fixed.
Success of cannulation | the day of intervention (Day 1)
  Comparison of cannulation success proportion at first attempt between the 2 groups. Cannulation at first attempt is a success if the needle is inserted at first attempt. A cannulation is defined as successful if the needle is inserted without resistance
Number of cannulation attempt | the day of intervention (Day 1)
  Comparison of the number of attempt before cannulation success in between the 2 groups. Conversion to ultrasound guidance in the anatomical guidance group will be taken into account.
Number of puncture attempt | day of intervention (Day 1)
  Comparison of the total number of puncture between the 2 groups. A puncture test is defined as the passage of the needle without changing direction or without new movement in depth. Each needle withdrawal, followed by a new movement to deep planes or redirection of the needle is regarded as a new test, with or without skin puncture. The number of tests will be evaluated by an observer.

CONTACTS AND LOCATIONS:
Overall Officials: Aurelie MAZAUD, MD, Principal Investigator — Department of intensive care unit, Hospital Edouard Herriot- Hospices Civils de Lyon
Locations (1):
- Department of intensive care unit, Hospital Edouard Herriot- Hospices Civils de Lyon, 5 Place d'Arsonval, Lyon, France

REFERENCES:
- [Result] Lazaar S, Mazaud A, Delsuc C, Durand M, Delwarde B, Debord S, Hengy B, Marcotte G, Floccard B, Dailler F, Chirossel P, Bureau-Du-Colombier P, Berthiller J, Rimmele T. Ultrasound guidance for urgent arterial and venous catheterisation: randomised controlled study. Br J Anaesth. 2021 Dec;127(6):871-878. doi: 10.1016/j.bja.2021.07.023. Epub 2021 Sep 6. PMID 34503827